CLINICAL TRIAL: NCT03811249
Title: A Prospective, Multicenter Clinical Trial of the VisAbility™ Micro Insert System for the Improvement of Near Visual Acuity in Presbyopic Subjects - Long Term Follow-up
Brief Title: Long Term Follow-up of the VisAbility™ Micro Insert System for Presbyopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Refocus Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIS-2014-5YR
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Presbyopia
Keywords: Near Vision; Reading Vision; Reading Glasses; Reading; Readers; Presbyopic
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Intervention Model Description: A non-randomized single group design. All subjects who were implanted with the VisAbility™ Micro Insert (360 subjects) will be invited to participate. Actual sample size will be determined at the completion of enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implantation-Non-randomized (Experimental): Subjects that previously participated in the VIS-2014 clinical trial that had VisAbility™ Micro Inserts surgically implanted in the eye(s) will be followed prospectively for an additional 36 month period to measure long term safety and effectiveness outcomes.
  Interventions: Device: VisAbility™ Micro Insert

INTERVENTIONS:
Device: VisAbility™ Micro Insert — No (new) intervention will be administered during the course of this long term follow-up study. Subjects that previously participated in the VIS-2014 clinical trial that had VisAbility™ Micro Inserts surgically implanted in the eye(s) will be followed prospectively.

SUMMARY:
The objective of this study is to obtain an additional 36 months of safety and effectiveness data from all subjects who were implanted with the VisAbility™ Micro Insert in the VIS-2014 clinical trial.

DETAILED DESCRIPTION:
VIS-2014-5YR is a multicenter, observational study to evaluate the long-term safety of the VisAbility™ Micro Inserts in subjects who were implanted with the VisAbility™ Micro Insert in the VIS-2014 clinical trial. Study subjects will be examined at 36, 48, and 60 months post-operatively (based on the anniversary of their first VisAbility™ surgery) with no planned interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were implanted with the VisAbility™ Micro Insert in Protocol VIS-2014

Exclusion Criteria:

* N/A

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schanzlin, Dr, Principal Investigator — Chief Medical Officer
Locations (13):
- United States (13):
  - Coastal Vision, Orange, California
  - Gordon Schanzlin New Vision Institute, San Diego, California
  - Aloha Laser Vision, Honolulu, Hawaii
  - The Midwest Center for Sight, Des Plaines, Illinois
  - Eye Surgeons Of Indiana PC, Indianapolis, Indiana
  - Eye Care Institute, Louisville, Kentucky
  - Chu Vision Institute, Bloomington, Minnesota
  - South Shore Eye Care LLP, Wantagh, New York
  - Physicians Protocol, Greensboro, North Carolina
  - Comprehensive EyeCare of Central Ohio, Westerville, Ohio
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Key Whitman Eye Center, Dallas, Texas
  - Braverman-Terry-Oei-Eye Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.refocus-group.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 13 clinical sites and consisted of contacting all subjects who were implanted or explanted in Protocol VIS-2014, a prospective multicenter clinical trial of the VisAbility Micro Insert System. If inclusion criteria was met, subjects who wished to participate provided written informed consent and were enrolled in this VIS-2014-5YR multicenter observational long-term study.
Pre-assignment Details: Per the protocol, primary and secondary safety outcome analysis was performed on all eyes of enrolled subjects that were implanted or explanted with the VisAbility Micro Insert System in the VIS-2014 clinical study. Secondary effectiveness analysis was performed on the primary eye of only those subjects who were bilaterally implanted (with all eight implants in place) in the VIS-2014 study, therefore, the primary eye is the unit of analysis for the secondary effectiveness outcome.
Units Other Than Participants: Eye
Groups:
- Implantation or Explantation Safety Cohort: Subjects that previously participated in the VIS-2014 clinical trial that had VisAbility™ Micro Inserts surgically implanted or explanted in the eye(s) will be followed prospectively for an additional 36 month period to measure long term safety outcomes.
  VisAbility™ Micro Insert: No (new) intervention will be administered during the course of this long term follow-up study. Subjects that previously participated in the VIS-2014 clinical trial that had VisAbility™ Micro Inserts surgically implanted or explanted in the eye(s) will be followed prospectively.
Period: Overall Study
Arm/Group | Implantation or Explantation Safety Cohort
Started | 287; 565 Eye (Subjects were allowed to enroll during any phase of the long-term follow-up study through the closure of the 60 month window. Due to the timing of study initiation, many subjects had already passed the 36 month window by the time enrollment ensued.)
Completed | 219; 433 Eye
Not Completed | 68; 132 Eye
Not completed — Withdrawal by Subject | 44
Not completed — Missed Visit | 24

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (eyes) | 565
Age, Continuous [Mean (Full Range); unit: years] | 51.7 [45 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 260
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 16
  Black or African American | 13
  Caucasian | 243
  Native Hawaiian or Other Pacific Islander | 4
  Other | 11
Dominant Eye [Number; unit: participants]
  OD | 190
  OS | 97
Distance Corrected Near Visual Acuity (DCNVA-Logarithm of the Minimum Angle of Resolution(LogMAR)))) [Mean (Standard Deviation); unit: LogMAR] — Preoperative LogMAR Distance Corrected Near Visual Acuity measured at 40cm. This represents the near visual acuity with the distance refractive correction in front of the eye.
  LogMAR | 0.496 (0.083)
Uncorrected Near Visual Acuity ((UCNVA-Logarithm of the Minimum Angle of Resolution (LogMAR)) [Mean (Standard Deviation); unit: LogMAR] — Preoperative LogMAR Uncorrected Near Visual Acuity (UCNVA)at 40cm. This represents the near visual acuity without the distance refraction correction.
  LogMAR | 0.525 (0.084)
Bilateral Uncorrected Intermediate Visual Acuity (UCIVA LogMAR) [Mean (Standard Deviation); unit: LogMAR] — Preoperative LogMAR Bilateral (OU) Uncorrected Intermediate Visual Acuity (66cm). This represents the visual acuity at 66cm while both eyes are viewing without any distance refraction correction in place.
  LogMAR | 0.335 (0.151)
Uncorrected Distance Visual Acuity (UCDVA LogMAR) [Mean (Standard Deviation); unit: LogMAR] — Preoperative LogMAR uncorrected distance visual acuity (6m). This represents the vision in each eye while looking at distance (6 meters) without the distance refractive correction in place.
  LogMAR | -0.011 (0.091)
Best Corrected Distance Visual Acuity (BCDVA-LogMAR) [Mean (Standard Deviation); unit: LogMAR] — Preoperative LogMAR Best Corrected Distance Visual Acuity (6m). This represents the distance visual acuity in each eye with the distance refraction correction in place.
  LogMAR | -0.072 (0.065)
Manifest Refraction Spherical Equivalent (MRSE-Diopters)) [Mean (Standard Deviation); unit: Diopters] — Preoperative Manifest Refraction Spherical Equivalent in Diopters
  Diopters | 0.129 (0.261)
Near Addition (D) [Mean (Standard Deviation); unit: Diopter] — Preoperative Near Addition over the distance refractive correction in Diopters required to see 20/20
  Diopter | 1.617 (0.306)
Intraocular Pressure (IOP-mmHg) [Mean (Standard Deviation); unit: mmHg] — Preoperative Intraocular Pressure in mmHg
  mmHg | 14.7 (2.6)
Maximum Pupil Size (mm) [Mean (Standard Deviation); unit: millimeters] — Preoperative maximum (scotopic=dim lighting of dark adapted eyes) pupil size in mm
  millimeters | 5.53 (0.79)
Minimum Pupil Size (mm) [Mean (Standard Deviation); unit: millimeters] — Preoperative minimum (photopic) pupil size in mm
  millimeters | 3.18 (0.56)
Astigmatism (D) [Mean (Standard Deviation); unit: Diopters] — Preopeartive Refractive Astigmatism in Diopters
  Diopters | -0.285 (0.289)
Cycloplegic Spherical Equivalent (D) [Mean (Standard Deviation); unit: Diopters] — Preoperative Spherical Equivalent after cycloplegia in Diopters
  Diopters | 0.222 (0.304)
Corneal Keratometry [Mean (Standard Deviation); unit: Diopters] — Preoperative Mean Corneal Keratometry (K1+K2)/2 in Diopters
  Diopters | 43.664 (1.371)
Scleral Thickness [Mean (Standard Deviation); unit: microns] — Preoperative Scleral Thickness measured 3.5mm from limbus in the superior temporal quadrant in units of Microns
  microns | 572.6 (44.2)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Measure - Partial or Complete Explantation
Description: Partial explantation (surgical removal of 1-3 Micro Inserts per eye), or complete explantation (surgical removal of all 4 Micro inserts per eye), and reason(s). Safety measure will be recorded if the event occurs.
Time Frame: From date of VIS-2014-5YR enrollment until the date of study withdrawal or study completion, whichever comes first, assessed up to 60 months post-surgery.
Population: All implanted or explanted eyes in the VIS-2014 clinical study who were subsequently enrolled in the VIS-2014-5YR long term study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes
  Partial Explant | 2
  Complete Explant | 4

2. Primary Outcome: Primary Safety Measure - Anterior Segment Ischemia
Description: Anterior Segment Ischemia (decreased blood perfusion to the anterior segment of the eye (Grades 2 - 4--the higher the grade, the worse the outcome).
  Grade 2 is decreased pupil reactivity (<25% of Percent Constriction using Neuroptics Pupillometry) Grade 3 is decreased pupil reactivity, plus anterior chamber reaction of Grade 2 cell and/or flare as assessed via biomicrosope examination Grade 4 is decreased pupil reactivity, plus anterior chamber reaction of Grade 2 cell and/or flare, plus corneal edema (Grade 3 with Striate Keratopathy) as assessed via biomicroscope examination Safety measure will be recorded if the event occurs.
Time Frame: as for outcome 1
Population: All eyes that were previously implanted or explanted in the VIS-2014 clinical trial
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes | 0

3. Primary Outcome: Primary Safety Measure - Segment Exposure.
Description: Segment exposure due to conjunctival and/or scleral erosion as assessed via biomicroscopic examination. Safety measure will be recorded if the event occurs.
Time Frame: as for outcome 1
Population: All eyes implanted or explanted in the VIS-2014 clinical study.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes | 1

4. Primary Outcome: Primary Safety Measure -Participants With Serious Ocular and Serious Non-Ocular Adverse Events
Description: Rate of Individual Participants with Serious Ocular and Serious Non-Ocular Adverse Events (SAE's). Safety measure will be recorded if the event occurs.
Time Frame: as for outcome 1
Population: Subjects that were enrolled and implanted or explanted in the VIS-2014 clinical trial and subsequently enrolled in the VIS-2014-5YR long term study.
Measure: Count of Participants; unit: Participants
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Participants
  Participants with Ocular Serious Adverse Events | 0
  Participants with Non-Ocular Serious Adverse Events | 4
  Ischemic Stroke leading to Cortical Left Inferior Homonymous Hemianopsia | 1
  COVID-19 Infection | 1
  Hepatic Encephalopathy | 1
  Sepsis of Left Lower Leg leading to BKA and Coma | 1

5. Secondary Outcome: Secondary Safety Measure - Best Corrected Distance Visual Acuity (BCDVA) in Eyes Examined at 36, 48 and 60 Month Visits
Description: Best Corrected Distance Visual Acuity (BCDVA, which is distance visual acuity with the best distance refractive corretion in place) in all eyes seen at the 36 month postoperative visit, 48 month postoperative visit and 60 month postoperative visit will be measured and recorded.
Time Frame: From date of enrollment until the date of study withdrawal or study completion, whichever comes first, assessed up to 60 months post-surgery.
Population: BCDVA for all eyes that were implanted or explanted in the VIS-2014 and subseuqently enrolled in the VI-2014-5YR long term study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes
  Percentage of eyes achieving BCDVA of 20/20 or better at 36 months postoperative visit: number analyzed (Participants) | 186
  Percentage of eyes achieving BCDVA of 20/20 or better at 36 months postoperative visit: number analyzed (Eyes) | 368
  Percentage of eyes achieving BCDVA of 20/20 or better at 36 months postoperative visit | 363
  Percentage of eyes with BCDVA of 20/20 or better at 48 months postoperative: number analyzed (Participants) | 267
  Percentage of eyes with BCDVA of 20/20 or better at 48 months postoperative: number analyzed (Eyes) | 526
  Percentage of eyes with BCDVA of 20/20 or better at 48 months postoperative | 510
  Percentage of eyes achieving BCDVA of 20/20 or better at 60 months postoperative: number analyzed (Participants) | 219
  Percentage of eyes achieving BCDVA of 20/20 or better at 60 months postoperative: number analyzed (Eyes) | 433
  Percentage of eyes achieving BCDVA of 20/20 or better at 60 months postoperative | 330

6. Secondary Outcome: Secondary Safety Measure - Intraocular Pressure (IOP)
Description: IOP increase > 10 mm Hg over baseline or IOP > 30 mm Hg as measured via Goldmann applanation tonometry
Time Frame: From date of enrollment until the date of study withdrawal or study completion, whichever came first, assessed up to 60 months post-surgery.
Population: Safety Cohort Consists of all implanted or explanted eyes in the VIS-2014 who enrolled in the VIS-2014-5YR long term study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 36 month visit | 0
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 48 month visit: number analyzed (Participants) | 267
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 48 month visit: number analyzed (Eyes) | 526
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 48 month visit | 0
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 60 month visit: number analyzed (Participants) | 219
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 60 month visit: number analyzed (Eyes) | 433
  # of eyes with IOP <6mmHg, or >30mmHg, or an increase in IOP >10mmHg from baseline at 60 month visit | 0

7. Secondary Outcome: Secondary Safety Measure - Slit Lamp
Description: Slit Lamp findings in all eyes implanted or explanted during the VIS-2014 clinical study and subsequently enrolled in the VIS-2014-5YR
Time Frame: as for outcome 1
Population: Eyes implanted or explanted during the VIS-2014 clinical study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes
  Mild Superficial Punctate Keratitis | 11
  Corneal Abrasion | 0
  Corneal Edema | 0
  Corneal Endothelial Guttata more than rare | 0
  Mild Conjunctival Injection not noted preoperatively | 17
  Subconjunctival hemorrhage of 2 quadrants or less | 7
  Trace Conjunctival Edema | 2
  Conjunctival Cyst | 3
  Conjunctival Scar | 5
  Pyogenic Granuloma | 1
  Anterior Chamber Cell | 0
  Anterior Chamber Flare | 0
  Iris Atrophy | 2
  2 Grade change in Lens Opacity | 8

8. Secondary Outcome: Secondary Safety Measure - Fundus Exam
Description: Fundus exam findings (using binocular indirect ophthalmoscopy and/or the biomicroscope/slit lamp and a condensing lens) in all eyes implanted or explanted in the VIS-2014 clinical study and subsequently enrolled in the VIS-2014-5YR study
Time Frame: as for outcome 1
Population: Implanted or explanted eyes in the VIS-2014 clinical study subsequently enrolled in the VIS-2014-5YR study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Number analyzed (Eyes) | 565
Eyes
  Age Related Macular Degeneration | 2
  Longstanding Branch Retinal Vein Occlusion | 1
  Central Serous Retinopathy | 2
  Chorioretinal Scars | 2
  Choroidal Nevi | 7
  Cotton Wool Spots | 3
  Epiretinal Membranes | 2
  Lattice Degeneration | 5
  Microaneurysms | 1
  Optic Nerve Pallor 2ndary to stroke or neuropathy | 3
  Peripheral Retinal Degeneration | 2
  Presumed Ocular Histoplasmosis Syndrome (POHS) | 2
  Posterior Vitreous Detachment | 6
  REtinal Pigment Epithelium changes | 4
  Retinal Pigment Epithelial detachment | 1
  RPE hyperplasia 2ndary to laser treatment | 1

9. Secondary Outcome: Secondary Safety Measure - Number of Participants With Adverse Events
Description: Rate of Adverse Events (AE's) in all participants implanted or explanted during the VIS-2014 clinical study and subsequently enrolled in the VIS-2014-5YR study
Time Frame: as for outcome 1
Population: Subjects who were either implanted or explanted during the VIS-2014 clinical study and subsequently enrolled in the VIS-2014-5YR Long Term study
Measure: Count of Participants; unit: Participants
Arm/Group | Implantation or Explantation Safety Cohort
Number analyzed (Participants) | 287
Participants
  BCDVA loss greater than or equal to 2 lines | 4
  Lids and Lashes (Chalazion lid margin disease) | 3
  Dry Eye signs requring prescription | 2
  Conjunctival Cyst | 3
  Conjunctival Erosion | 1
  Subconjunctival hemorrhage (not associated with an explant, concomitant procedure, etc.) | 5
  Conjunctivitis (allergic, bacterial, viral) | 3
  Scleral Erosion | 0
  Persistent Pupil Abnormality | 0
  Anterior Segment Ischemia | 0
  Lens Opacity-2 grade change as compared to preoperative baseline | 7
  Glaucoma | 0
  Posterior Vitreous Detachment-new onset | 2
  Extruded, Misplaced or Missing Segments | 0
  Complete Explantation | 2
  Partial Explantation | 2
  Cataract Extraction | 2
  Other 2ndary Surgical Procedure (Clear Lens Exchange or PRK) | 3
  Central Serous Chorioretinopathy | 2
  Chemical Injury | 1
  Cotton Wool Spot | 1
  Dry Eye Symptoms requiring prescription medication | 2
  Epiretinal Membrane | 2
  Foreign Body Sensation | 1
  Lattice Degeneration | 1
  Non Proliferative Diabetic Retinopathy | 1
  Ocular Migraine | 1
  Pyogenic Granuloma | 1
  Recurrent Corneal Erosion | 1
  Trichiasis of single lash Right lower lid | 1

10. Secondary Outcome: Secondary Effectiveness Measure - Distance Corrected Near Visual Acuity--Effectiveness Cohort
Description: distance corrected near visual acuity of 20/40 or better in the primary eye of bilaterally implanted subjects (with all eight implants in place), as compared to baseline (VIS-2014).
Time Frame: as for outcome 1
Population: Primary eyes of subjects who were bilaterally implanted during the VIS-2014 clinical study, were subsequently enrolled in the VIS-2014-5YR study and have all 8 segments in place.
Measure: Count of Units; unit: Primary Eyes
Units Other Than Participants: Primary Eyes
Groups:
- Effectiveness Cohort: Subjects who were bilaterally implanted in the VIS-2014 clinical study and still have all 8 segments in place during the respective visit.
Arm/Group | Effectiveness Cohort
Number analyzed (Participants) | 262
Number analyzed (Primary Eyes) | 262
Primary Eyes
  Preopeartive DCNVA 20/40 or better | 2
  36 months DCNVA 20/40 or better: number analyzed (Primary Eyes) | 172
  36 months DCNVA 20/40 or better | 149
  48 months DCNVA 20/40 or better: number analyzed (Primary Eyes) | 242
  48 months DCNVA 20/40 or better | 212
  60 months DCNVA 20/40 or better: number analyzed (Primary Eyes) | 193
  60 months DCNVA 20/40 or better | 161

11. Secondary Outcome: Secondary Effectiveness Measure--Uncorrected Near Visual Acuity-Effectivness Cohort
Description: uncorrected near visual acuity of 20/40 or better in the primary eye of bilaterally implanted subjects (with all eight implants in place), as compared to baseline (VIS-2014).
Time Frame: as for outcome 1
Population: Number of primary eyes of bilaterally implanted subjects (with all 8 segments in place) present at each visit (preopeartive, 36, 48 and 60 months)
Measure: Count of Units; unit: Primary Eyes
Units Other Than Participants: Primary Eyes
Arm/Group | Effectiveness Cohort
Number analyzed (Participants) | 262
Number analyzed (Primary Eyes) | 262
Primary Eyes
  Primary Eye UCNVA 20/40 or better at baseline | 2
  Primary Eye UCNVA 20/40 or better at 36 months: number analyzed (Participants) | 172
  Primary Eye UCNVA 20/40 or better at 36 months: number analyzed (Primary Eyes) | 172
  Primary Eye UCNVA 20/40 or better at 36 months | 135
  Primary Eye UCNVA 20/40 or better at 48 months: number analyzed (Participants) | 242
  Primary Eye UCNVA 20/40 or better at 48 months: number analyzed (Primary Eyes) | 242
  Primary Eye UCNVA 20/40 or better at 48 months | 174
  Primary Eye UCNVA 20/40 or better at 60 months: number analyzed (Participants) | 193
  Primary Eye UCNVA 20/40 or better at 60 months: number analyzed (Primary Eyes) | 193
  Primary Eye UCNVA 20/40 or better at 60 months | 128

ADVERSE EVENTS:
Time Frame: From date of VIS-2014-5YR enrollment until the date of study withdrawal or study completion, whichever comes first, assessed up to 60 months post-surgery
Arm/Group | Implantation or Explantation Safety Cohort
All-Cause Mortality (participants affected / at risk) | 0/287
Serious Adverse Events (participants affected / at risk) | 4/287
Other Adverse Events (participants affected / at risk) | 46/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation or Explantation Safety Cohort (N=287)
Ischemic Stroke w/ 2ndary Cortical Left Inferior Homonymous Hemianopsia (Nervous system disorders) | 1 (1) — Non-Ocular Non-Device Related Serious Adverse Event
COVID-19 Infection (Infections and infestations) | 1 (1) — Non-Ocular, Non-Device Related Serious Adverse Event
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 (1) — Non-Ocular Non-Device Related Serious Adverse Event
Sepsis of the Left Lower Leg leading to BKA and Coma (Infections and infestations) | 1 (1) — Non-Ocular Non-Device related Serious Adverse Event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implantation or Explantation Safety Cohort (N=287)
Decrease in BCDVA of greater than or equal to 2 lines (Eye disorders) | 4 (5) — Decrease in BCDVA of greater than or equal to 2 lines
Chalazion/Lid Margin Disease (Eye disorders) | 3 (4) — Chalazion, or onset of or worsening to severe, clinically signficant lid margin disease
Dry Eye signs requiring prescription (Eye disorders) | 2 (4) — Dry Eye signs requiring prescription medication
Conjunctival Cyst (Eye disorders) | 3 (3) — Conjunctival Cyst
Conjunctival Erosion (Eye disorders) | 1 (1) — Conjunctival Erosion
Subconjunctival hemorrhage (Eye disorders) | 5 (6) — Subconjunctival hemorrhage not associated wtih an explant, concomitant procedure, etc.
Conjunctivitis (Eye disorders) | 3 (6) — Conjunctivitis (allergic, bacterial, or viral)
Lens Opacity (Eye disorders) | 7 (8) — Lens Opacity--2 grade change as compared to preoperative baseline
Posterior Vitreous Detachment (Eye disorders) | 2 (2) — Posterior Vitreous Detachment
Secondary Surgical Intervention-Complete Explant (Eye disorders) | 2 (4) — Explant of all 4 segments or all remaining segments from eye
Secondary Surgical Intervention-Partial Explant (Eye disorders) | 2 (2) — Individual or multiple segments removed with at least 1 remaining segment
Secondary Surgical Intervention-Cataract Extraction (Eye disorders) | 2 (3) — Cataract Extractiion
Other Surgical Intervention (Eye disorders) | 3 (5) — Other Surgical interventon--clear lens extraction, photorefractive keratectomy
Central Serous Chorioretinopathy (Eye disorders) | 2 (2) — Central Serous Chorioretinopathy
Chemical Injury (Injury, poisoning and procedural complications) | 1 (1) — non-devic, non-procedure related ocular chemical injury
cotton wool spot (Eye disorders) | 1 (1) — retinal finding associated with systemic hypertension
Dry Eye Symptoms requiring prescription medication (Eye disorders) | 4 (4) — Patient reports of dry eye symptoms despite no clinical signs of dry eye--prescription medication was prescribed
Epiretinal membrane (Eye disorders) | 2 (2) — Epiretinal membrane
Foreign Body Sensation (Eye disorders) | 1 (1) — Ocular Foreign Body Sensation
Lattice Degeneration (Eye disorders) | 2 (2) — Lattice Degeneration
Non-Proliferative Diabetic Retinopathy (Endocrine disorders) | 1 (1) — Non-device related finding associated with systemic diabetes
Ocular Migraine (Vascular disorders) | 1 (1) — Ocular Migraine
Pyogenic Granuloma (Eye disorders) | 1 (1) — Pyogenic Granuloma
Recurrent Corneal Erosion (Eye disorders) | 1 (1) — Injury related recurrent corneal erosion, not device or procedure related
Trichiasis of single lash right lower lid (Eye disorders) | 1 (1) — Not device/procedure related

LIMITATIONS AND CAVEATS:
Delay in VIS-2014-5YR approval and initiation resulted in some of the participants falling outside the 36 month window at the time of study commencement.

COVID shutdowns affected study accountability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor encourages publication and presentation of the safety and effectiveness results upon completion of the study. Per the established investigator agreement, the Principal Investigators will work with the Sponsor, in good faith, to ensure all confidential and proprietary informaton is redacted.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03811249/Prot_SAP_000.pdf